CLINICAL TRIAL: NCT06877286
Title: The Relationship Between EPO Resistance and Sirtuin-1 Levels in Hemodialysis Patients.
Brief Title: Low Sirtuin-1 Levels Are Linked to Erythropoietin Resistance in Hemodialysis Patients.
Status: Completed | Type: Observational
Sponsor: Cuma Bulent Gul (Other)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Cuma Bulent Gul, Professor, Uludag University
Organization: Uludag University (Other)
Other Study IDs: SIRT1-EPO-2020; 2011-KAEK-25 2020/07-06 (Other: Bursa Yuksek Ihtisas Hospital Ethics Committee)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Anemia in End Stage Renal Disease; Erythropoietin
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples were retained at -80°C for SIRT1 analysis and subsequently discarded after analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemodialysis Patients: Patients with erythropoietin resistance undergoing hemodialysis.
  Interventions: Diagnostic Test: Sirtuin-1 Level Measurement

INTERVENTIONS:
Diagnostic Test: Sirtuin-1 Level Measurement — Measurement of serum Sirtuin-1 levels using ELISA in hemodialysis patients to evaluate the relationship between Sirtuin-1 levels and erythropoietin resistance

SUMMARY:
This study investigates the relationship between Sirtuin-1 (SIRT1) levels and erythropoietin resistance in hemodialysis patients. The study aims to determine whether low SIRT1 levels contribute to EPO resistance and to explore the potential mechanisms involved. Blood samples and clinical data from hemodialysis patients will be analyzed to evaluate this relationship.

DETAILED DESCRIPTION:
This study explores the association between Sirtuin-1 (SIRT1) levels and erythropoietin resistance in hemodialysis patients. Erythropoiesis-stimulating agents (ESAs) are commonly used to treat anemia in chronic kidney disease (CKD) patients undergoing hemodialysis. However, a significant proportion of patients exhibit hyporesponsiveness to ESAs, leading to suboptimal anemia management. SIRT1, a nicotinamide adenine dinucleotide (NAD+)-dependent histone deacetylase, regulates hypoxia and iron metabolism by modulating the activity of hypoxia-inducible factor 1α (HIF-1α). Lower SIRT1 levels may impair HIF-1α activity and contribute to reduced erythropoietin (EPO) responsiveness.

In this multicentric cross-sectional cohort study, 391 adult hemodialysis patients from provincial dialysis clinics in Bursa, Turkey, were enrolled between August 2020 and March 2021. ESA responsiveness was assessed using the Erythropoietin Resistance Index (ERI), calculated as the weekly weight-adjusted ESA dose divided by hemoglobin concentration. Serum SIRT1 levels were measured using a human SIRT1 ELISA kit.

The study aims to determine whether low SIRT1 levels are independently associated with higher ERI scores and to identify other clinical and biochemical parameters influencing ESA responsiveness. Multiple regression and correlation analyses will be performed to evaluate the relationship between SIRT1 levels, ERI scores, ferritin levels, and other clinical factors. Logistic regression will also be conducted to explore whether SIRT1 is an independent predictor of high ERI scores (≥50th percentile).

The findings from this study may provide new insights into the molecular mechanisms underlying ESA resistance and highlight the potential role of SIRT1 as a target for improving anemia management in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Receiving hemodialysis
* Availability of laboratory data to calculate ERI

Exclusion Criteria:

* Autosomal polycystic kidney disease
* Malignancies
* Infectious diseases
* Chronic rheumatological disorders
* Vitamin B12 or folic acid deficiency
* CRP levels ≥ 5 mg/L
* PTH levels ≥ 300 pg/dL
* Inadequate hemodialysis (Kt/Vurea < 1.2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) undergoing hemodialysis in provincial hemodialysis clinics in Bursa, Turkey, between August 2020 and March 2021. Eligible patients had available laboratory data to calculate the Erythropoietin Resistance Index (ERI). Patients with certain comorbidities, such as malignancies, infectious diseases, chronic rheumatological disorders, and vitamin deficiencies, were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Sirtuin-1 levels | Measured at baseline (initial blood sample)
  Measurement of serum Sirtuin-1 levels using ELISA to evaluate its association with erythropoietin resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag University Medical School, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality and data privacy regulations.